CLINICAL TRIAL: NCT04343612
Title: The Effects of Different Montages of Transcranial Direct Current Stimulation on Tongue Strength in Healthy Subjects
Brief Title: Different Montages of Transcranial Direct Current Stimulation Tongue Strength
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Bornheim Stephen, Assistant Professor, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-93
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: tDCS; IOPI; Tongue Strength; Healthy
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: 4 groups, each group receives one of three treatments or the sham treatment. Double-blinded, sham controlled, crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Everyone is blinded, codes are selected by a third party not involved in any step of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anodal (Experimental): Anode placer over the affected primary motor cortex, cathode over contralateral supra orbital area. 2 mA, 20min stimulation
  Interventions: Device: Transcranial Direct Current Stimulation
- Bilateral (Experimental): Anode placer over the affected primary motor cortex, cathode over unaffected motor cortex. 2 mA, 20min stimulation
  Interventions: Device: Transcranial Direct Current Stimulation
- Cathodal (Experimental): Cathode placer over the unaffected primary motor cortex, anode over contralateral supra orbital area. 2 mA, 20min stimulation
  Interventions: Device: Transcranial Direct Current Stimulation
- Placebo (Placebo Comparator): anode montage but current is ramped up over 15 secondes, then ramped down. 2 mA, 20min stimulation
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Subjects received a micro-current through their scalp to induce cortical and subcortical changes
  Other Names: tDCS

SUMMARY:
20 healthy subjects will be split into 4 groups. Each group will receive one of the following tDCS montages : anodal, bilateral, cathodal or placebo Subjects will receive 2mA for 20 mins of their attributed tDCS. The evaluation is a maximal strength test measured with the IOPI and will take place prior to, immediately following and 30 minutes after stimulation

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* One Yes on the medium and high risk sections of the TSST (Bornheim et al.,2019)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Change Tongue Maximal Strength | Baseline, immediately after, and 30 minutes after tDCS
  1 RM of tongue strength, measured using the IOPI device

CONTACTS AND LOCATIONS:
Locations (1):
- Liege Univeristy, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bornheim S, Croisier JL, Maquet P, Kaux JF. Proposal of a New Transcranial Direct Current Stimulation Safety Screening Tool. Am J Phys Med Rehabil. 2019 Jul;98(7):e77-e78. doi: 10.1097/PHM.0000000000001096. No abstract available. PMID 30431445